CLINICAL TRIAL: NCT06783972
Title: The Effect of Touching the Fetal Head of the Pregnant on the Duration of the Second Stage of Labor and the Mother-Baby Interaction During the Perineal Crowning Phase
Brief Title: The Effect of Touching the Fetal Head During the Perineal Crowning Phase
Acronym: Touching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Dilek Mamik Aktay, Midwife, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ethics Committee Number 942
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-01

CONDITIONS: The Effect of Touching the Fetal Head of the Pregnant on the Duration of the Second Stage of Labor
Keywords: midwifery; vaginal birth; touching
MeSH Terms: interventions — Touch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (No Intervention): Routine labor monitoring
- Group 2 (Experimental): fetal head touching practice
  Interventions: Behavioral: Touching

INTERVENTIONS:
Behavioral: Touching — In the second stage of birth, when the baby's head crowns, the mother is allowed to touch the baby's head as much as she wants and with as many fingers as she wants.
  Arms: Group 2

SUMMARY:
In this study, it is planned to shorten the second stage of labor by touching the fetal head during the second stage of labor. It is thought that touching will also have positive effects on the mother and the newborn. The fact that touching the fetal head is a cost-free and easily applicable action is a different and strong aspect from other studies. This research study that we have planned is quite meaningful in terms of ensuring a comfortable postpartum period within the scope of mother and baby-friendly practices that our Ministry emphasizes.

ELIGIBILITY:
Inclusion Criteria:

* Not to have obstetric risk,
* To be primiparous,
* To be 37W and above pregnant,
* To carry a live fetus,
* To be mentally healthy,
* To be able to communicate,
* To be literate,
* To have no systemic disease,
* To not use medication for any reason,
* To have no addiction, no movement restriction

Exclusion Criteria:

* Leaving the study before it is completed

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 68 (Actual)
Dates: Start 2025-01-19 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Mother-Baby Interaction | This scale was applied on the 1st and 2nd day after birth.
  The research output will be evaluated with the Mother-Infant Interaction Scale. This scale is a three-point Likert-type scale from positive to negative, aiming to determine the mother's responses, reactions and closeness to her baby in the early postpartum period. There are 5 behavioral classifications for the mother in each scale. These are grouped as; Sensitivity for the baby, Touching/holding, Eye-to-eye and face-to-face communication, Providing adequate care, Expressing feelings. In order to obtain a full score on the scale; the item that gives the best description from each of the five behavioral categories is marked. Each item in the five behavioral categories is grouped by giving "2,1,0" points. At the end of the observation, each category is scored and a total score is obtained. The scale is applied by observing the behaviors of the mother and her baby during the first contact and the 2nd day after birth. With the scores obtained, the midwife determines the

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data security

REFERENCES:
- [Result] Feldman R, Singer M, Zagoory O. Touch attenuates infants' physiological reactivity to stress. Dev Sci. 2010 Mar;13(2):271-8. doi: 10.1111/j.1467-7687.2009.00890.x. PMID 20136923
- [Result] Goldstein P, Weissman-Fogel I, Shamay-Tsoory SG. The role of touch in regulating inter-partner physiological coupling during empathy for pain. Sci Rep. 2017 Jun 12;7(1):3252. doi: 10.1038/s41598-017-03627-7. PMID 28607375
- [Result] Hertenstein MJ, Keltner D, App B, Bulleit BA, Jaskolka AR. Touch communicates distinct emotions. Emotion. 2006 Aug;6(3):528-33. doi: 10.1037/1528-3542.6.3.528. PMID 16938094
- [Result] Sehlstedt I, Ignell H, Backlund Wasling H, Ackerley R, Olausson H, Croy I. Gentle touch perception across the lifespan. Psychol Aging. 2016 Mar;31(2):176-84. doi: 10.1037/pag0000074. PMID 26950227
- [Result] Tang Y, Benusiglio D, Lefevre A, Hilfiger L, Althammer F, Bludau A, Hagiwara D, Baudon A, Darbon P, Schimmer J, Kirchner MK, Roy RK, Wang S, Eliava M, Wagner S, Oberhuber M, Conzelmann KK, Schwarz M, Stern JE, Leng G, Neumann ID, Charlet A, Grinevich V. Social touch promotes interfemale communication via activation of parvocellular oxytocin neurons. Nat Neurosci. 2020 Sep;23(9):1125-1137. doi: 10.1038/s41593-020-0674-y. Epub 2020 Jul 27. PMID 32719563
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32719563/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26950227/